CLINICAL TRIAL: NCT02638779
Title: REAnimation Low Immune Status Markers
Acronym: REALISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Bioaster (Other); BioMérieux (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL15_0379; 2015-A01293-46 (Other: ID-RCB)
Record Dates: First submitted 2015-12-18; First posted 2015-12-23 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Septic Shock; Severe Trauma; Severe Burn; Major Surgery
Keywords: Septic shock; severe trauma; severe burn; major surgery; immunosuppression; Healthcare-Associated Infections
MeSH Terms: conditions — Shock, Septic; Wounds and Injuries; Burns; Cross Infection | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood sampling (Experimental): Blood sampling will be performed in all patients and healthy volunteers
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Specific Blood sampling will be performed in patients and healthy volunteers

SUMMARY:
The fact that sepsis disrupts immune system homeostasis by inducing an initial cytokine storm, that participates to occurrence of organ failures and early death, followed by a compensatory anti-inflammatory response leading to immunosuppression, is now well established. This immunomodulating response results in a higher risk of secondary infections and is associated to 2/3 of deaths related to septic shocks. Follow up of patients' immune status with time is crucial to guide therapy management. Objective of REALISM project is to demonstrate existence of this immunosuppression phase, by providing strong epidemiologic data for septic shock patients, but also by extension to other situations of inflammatory aggressions like severe severe trauma or burns, or major surgery. This project will provide tools to predict occurrence of secondary infections and guide patient management by comparing innovating immunomonitoring tools to reference tests non already adapted to a routine patient management.

Targeted populations are adult patients hospitalized for septic shock, severe trauma (including severe burn) or major surgery and healthy volunteers, whom blood samples will serve to validate reference intervals of the two reference tests.

ELIGIBILITY:
Inclusion criteria for patients

* Patient or next of kin having been informed of the conditions of the study and having signed the informed consent form
* Patient hospitalized for :

  * Septic shock
  * Severe trauma (including severe burn)
  * Major surgery

Inclusion criteria for healthy volunteers

* Normal clinical examination
* Signed informed consent form
* Person with social security insurance

Exclusion criteria for patients

* Patient with severe neutropenia (neutrophil count <0.5 g/l)
* Patients receiving immunosuppressive therapy
* Patients receiving corticosteroids (IV or Per os)
* Use of therapeutic antibodies
* Hematological disease under treatment, or treated within 5 years before inclusion
* End of chemotherapy within the 6 months prior to inclusion
* Patient with innate or acquired immune deficiency (for example severe combined immunodeficiency, HIV or AIDS, any stage)
* Patients for whom a care limitation was pronounced at time of enrolment
* Anticipated length of stay before discharge from the ICU is estimated at less than 48 hours
* Participation in an intervention study
* Extra-corporeal circulation in the month preceding inclusion in case of cardiac surgery
* Pregnant or breastfeeding women
* Patient with no social security insurance, with restricted liberty or under legal protection

Exclusion criteria for healthy volunteers

* Person with an infectious syndrome during the last 90 days
* Extreme physical stress within the last week
* Person having received within the last 90 days, a treatment based on

  * Antivirals
  * Antibiotics
  * Antiparasitics
  * Antifungics
* Person having received within the last 15 days, a treatment based on non-steroidal anti-inflammatory drugs (NSAIDs)
* Person having received within the last 24 months, a treatment based on

  * Immunosuppressive therapy
  * Corticosteroids (IV or Per os)
  * Therapeutic antibodies
  * Chemotherapy
* History of :

  * innate or acquired immune deficiency
  * Hematological disease
  * Solid tumor
  * Severe chronic disease
  * Surgery or hospitalization within the last 2 years
  * Pregnancy within the last year
* Participation to a phase I clinical assay during the last year
* Pregnant or breastfeeding women
* Person with restricted liberty or under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
Percentage of patients meeting the definition of of injury-induced-immunosuppression | Up to 2 months after injury
  The immunosuppression status will be determined from two immunological reference tests: (1) lymphocyte proliferation in response to ex vivo T cell stimulation (adaptive immunity) (Poujol et al., 2014) and (2) the production of tumor necrosis factor (TNF) by monocytes in response to ex vivo stimulation by lipopolysaccharide (LPS) (innate immunity) (Duffy et al., 2014). The values measured will be defined as normal or abnormal, depending on whether they are within reference intervals (RI) derived from an independent set of healthy volunteers. For this purpose, the definition of immunosuppression will be: an abnormal result in at least one of the two "reference" tests (outside the reference intervals defining normal values), and on at least two consecutive samples. The same reference test must be abnormal in two successive samples examined for the patient to be considered immunosuppressed.

SECONDARY OUTCOMES:
Proportion of patients with a deficiency of the innate or adaptive immunity | Up to 2 months after injury
  Intensity of the innate immune deficiency will be measured using the production of TNF by monocytes in response to ex vivo stimulation by LPS (Duffy et al., 2014). Intensity of the adaptive immune deficiency will be measured using the lymphocyte proliferation in response to ex vivo T cell stimulation (Poujol et al., 2014). The values measured will be defined as normal or abnormal, depending on whether they are within reference intervals derived from an independent set of healthy volunteers. We will describe for all groups of patients:
  * The proportion of patients with a deficiency of the innate immunity, defined by an abnormal TNF secretion test result after LPS stimulation, for at least two consecutive samples.
  * The proportion of patients with a deficiency of the adaptive immunity, defined by an abnormal lymphocyte proliferation, for at least two consecutive samples.
  * The proportion of patients with at least one abnormal test on Days 1, 3-4, 5-7, 13/18, 26/36 and 52/68
Comparison of performance of the reference tests and new biomarkers for the diagnosis of immunosuppression | Up to one week after injury
  Reference tests being non-standardized and cumbersome to implement, and time to results being incompatible with clinical practice, the use of simpler and quicker tests, based on the use of new biomarkers, would allow the individualization of patient management based on the patient's immune status. One of the secondary objectives is to evaluate the performance of new biomarkers compared to the two reference tests to diagnose immunosuppression. Different types of markers and tests will be evaluated: Viral reactivation markers, host-response markers, immune functional assays, immunophenotyping.
Correlation between the immunosuppression status and the incidence of healthcare-associated infections | Up to 28 days after injury
  To evaluate the association between the immunosuppression status as defined in primary objective and the occurrence of secondary infections related to healthcare, the association of the immunosuppression status upon the occurrence of secondary infection will be examined first, and secondly any possible association between the levels of each of the reference tests and the occurrence of secondary infections will be characterized. In this analysis, a secondary infection related to healthcare will be defined as an infection occurring after inclusion in the study, between inclusion and day 28.
Correlation between immunosuppression and mortality | Up to 90 days after injury
  We will examine the association between immunosuppression (as defined in the primary objective) and in-hospital mortality. Association will be evaluated par measuring occurrence of mortality at days 14, 28, 60 and 90, in the different groups.
Comparison of immune status before and after surgery in the population of surgical patients | Up to 2 months after surgery
  The possibility of taking a sample before surgical stress should allow measurements of the impact of the procedure on the host response, and especially on any subsequent onset of immunosuppression. Oncological pathologies and treatments implemented prior to surgery may also be associated with immunosuppression, and for this reason patients hospitalized for cancer surgery will be compared to those hospitalized for vascular surgery. Impact of surgery on immunosuppression will be measured by comparing immune status as defined by the reference tests, in the population of surgical patients before and after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie Réanimation - Hôpital Edouard Herriot, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rol ML, Venet F, Rimmele T, Moucadel V, Cortez P, Quemeneur L, Gardiner D, Griffiths A, Pachot A, Textoris J, Monneret G; REALISM study group. The REAnimation Low Immune Status Markers (REALISM) project: a protocol for broad characterisation and follow-up of injury-induced immunosuppression in intensive care unit (ICU) critically ill patients. BMJ Open. 2017 Jun 21;7(6):e015734. doi: 10.1136/bmjopen-2016-015734. PMID 28637738
- [Result] Venet F, Textoris J, Blein S, Rol ML, Bodinier M, Canard B, Cortez P, Meunier B, Tan LK, Tipple C, Quemeneur L, Reynier F, Leissner P, Vedrine C, Bouffard Y, Delwarde B, Martin O, Girardot T, Truc C, Griffiths AD, Moucadel V, Pachot A, Monneret G, Rimmele T; REALISM study group. Immune Profiling Demonstrates a Common Immune Signature of Delayed Acquired Immunodeficiency in Patients With Various Etiologies of Severe Injury. Crit Care Med. 2022 Apr 1;50(4):565-575. doi: 10.1097/CCM.0000000000005270. PMID 34534131
- [Result] Mallet F, Diouf L, Meunier B, Perret M, Reynier F, Leissner P, Quemeneur L, Griffiths AD, Moucadel V, Pachot A, Venet F, Monneret G, Lepape A, Rimmele T, Tan LK, Brengel-Pesce K, Textoris J. Herpes DNAemia and TTV Viraemia in Intensive Care Unit Critically Ill Patients: A Single-Centre Prospective Longitudinal Study. Front Immunol. 2021 Nov 2;12:698808. doi: 10.3389/fimmu.2021.698808. eCollection 2021. PMID 34795661
- [Result] Peronnet E, Blein S, Venet F, Cerrato E, Fleurie A, Llitjos JF, Kreitmann L, Terraz G, Conti F, Gossez M, Rimmele T, Textoris J, Lukaszewicz AC, Brengel-Pesce K, Monneret G; REAnimation Low Immune Status Marker (REALISM) Study Group. Immune Profiling Panel Gene Set Identifies Critically Ill Patients With Low Monocyte Human Leukocyte Antigen-DR Expression: Preliminary Results From the REAnimation Low Immune Status Marker (REALISM) Study. Crit Care Med. 2023 Jun 1;51(6):808-816. doi: 10.1097/CCM.0000000000005832. Epub 2023 Mar 14. PMID 36917594
- [Derived] Bodinier M, Peronnet E, Brengel-Pesce K, Conti F, Rimmele T, Textoris J, Vedrine C, Quemeneur L, Griffiths AD, Tan LK, Venet F, Maucort-Boulch D, Monneret G; REALISM study group. Monocyte Trajectories Endotypes Are Associated With Worsening in Septic Patients. Front Immunol. 2021 Nov 29;12:795052. doi: 10.3389/fimmu.2021.795052. eCollection 2021. PMID 34912347